CLINICAL TRIAL: NCT06240923
Title: "Three Dimensional Assessment of Maxillary Molars Following Distalization Using Two Different Approaches"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Gihan Mohamed Anwar Mohamed Khattab, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORD 16-6M
Record Dates: First submitted 2023-12-12; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Malocclusion, Angle Class II
Keywords: Dental malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II; Malocclusion

STUDY DESIGN:
Intervention Model Description: A sample size of 24 maxillary dental distalizing sites were selected and divided into two groups twelve in each:
  Group 1: Single coil spring. Group 2: Double coil spring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Single coil spring (Experimental): A single open coil spring was inserted between the maxillary second premolar and the maxillary first molar with a distalizing force 300 gm.
  Interventions: Device: Maxillary molars distalization
- Group 2: Double coil spring (Experimental): Two open coil springs were inserted. The first coil spring was inserted between the maxillary second premolar and the maxillary first molar with a distalization force 300gm, and the second coil spring was inserted between the maxillary first and maxillary second molar with a distalization force 200 gm.
  Interventions: Device: Maxillary molars distalization

INTERVENTIONS:
Device: Maxillary molars distalization — Maxillary molars distalization by using a nickel titanium open coil spring as an posterior displacement device.
  Other Names: Posterior displacement of maxillary molars

SUMMARY:
The goal of this controlled clinical trial is to compare the effects of two distalization methods supported by inter-radicular mini-screw for maxillary molars distalization in 20 adult patients with skeletal class I or moderate skeletal class II malocclusion, dental class II molar relationship, and full permanent dentition. The participants were randomly selected according to inclusion / exclusion criteria from the outpatient clinic of the Department of Orthodontics and Dentofacial Orthopedics, Faculty of dentistry, Ain Shams University, Cairo, Egypt. Selectees age was ranging from 18 to 25 years old.

An informed consent has been signed by each patient before his / her enrollment in this study, where the aim , methodology, and possible complications were been clearly described in details. This research has been thoroughly reviewed by the Research Ethics Committee of the Faculty of dentistry, Ain Shams University.

DETAILED DESCRIPTION:
This study is a two-arm, parallel group, prospective randomized clinical trial with the allocation ratio of 1:1. The Consolidated Standards of Reporting Trials (CONSORT statement) were used as a guide for this study.

After reviewing the study protocol, the ethical committee at the Faculty of Dentistry, Ain-Shams University approved the study.

Before treatment was carried out, a detailed written Arabic consent was signed by all the subjects of both groups after full explanation of the aim of the study and the procedures.

This prospective clinical study was conducted on a total of 24 maxillary first molars.

No financial competing interests: This study was part of a Masters' degree in Orthodontics, Faculty of Dentistry, Ain-Shams University.

No financial conflicts of interest were declared. The study was self- funded by the principal investigator.

A sample size of 24 distalizing sites was selected and divided into two groups twelve each:

Group 1: Single coil spring. Group 2: Double coil spring.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects are free from any dental anomalies as well as periodontal and systemic diseases that may influence orthodontic treatment.
2. Adult patients with age ranging from 18 to 25 years.
3. Full permanent dentition with exclusion of third molars.
4. Both first and second maxillary molars are in occlusion.
5. Skeletal class I, mild or moderate skeletal class II malocclusion.
6. Full cusp or end to end class II molar relationship.
7. Mild to moderate crowding in the upper dental arch and / or increased overjet.
8. Normal or horizontal growth pattern.
9. Non-extraction treatment plan.

Exclusion Criteria:

1. Previous orthodontic treatment.
2. Treatment planning requiring orthognathic surgery.
3. Severe molar rotation.
4. Poor oral hygiene.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
The amount of maxillary molars distalization | 8-10 months
  Primary outcome of this study is to determine the amount of maxillary molars linear distal movement distance measured in millimeters.
The type of maxillary molars distalization | 8-10 months
  Molar tipping measured by the degree of the angle of tipping.

SECONDARY OUTCOMES:
Loss of anchorage | 8-10 months
  Anterior linear displacement of the premolars measured in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Noha I Abdelrahman, Assoc. Prof., Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF)

DOCUMENTS (3):
  • Study Protocol (2016-01-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT06240923/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT06240923/SAP_001.pdf
  • Informed Consent Form (2016-01-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT06240923/ICF_002.pdf